CLINICAL TRIAL: NCT05295095
Title: The Value of Positive Pressure Extubation in Reducing Postoperative Desaturation Episodes in Adults Undergoing Abdominal Surgery
Brief Title: Does Positive Pressure Extubation Reduce Postoperative Desaturation?
Acronym: EXTUBPOS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021_0433; 2021-A03064-37 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2022-02-21; First posted 2022-03-24 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-03

CONDITIONS: Extubation; Postoperative Complications; Lung Ultrasound Score
Keywords: positive pressure extubation; Postoperative Complications; lung ultrasound score
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Intervention Model Description: Single-center, prospective, controlled, parallel, randomized, single-blind study comparing the conventional extubation technique to two positive pressure extubation techniques
Who Masked: Participant
Masking Description: patients under anaesthesia at randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (No Intervention): Classical extubation technique : ETT was removed with continuous endotracheal suction
- VSPEP (Experimental): ETT was removed with APL valve set to 20cmH2O
  Interventions: Procedure: positive pressure during extubation procedure
- VSAIPEP (Experimental): ETT removed with ventilator parameters were set for PSV mode (inspiratory pressure of 10cmH2O and PEEP identical to that administered in the operating room
  Interventions: Procedure: positive pressure during extubation procedure

INTERVENTIONS:
Procedure: positive pressure during extubation procedure — positive pressure during extubation procedure
  Arms: VSAIPEP; VSPEP

SUMMARY:
Single-center, prospective, controlled, parallel, randomized, single-blind study comparing the conventional extubation technique to two positive pressure extubation techniques on postoperative desaturations

DETAILED DESCRIPTION:
Study realise on university hospital on Lille in France. Patients inclusion is prospective and randomised in three groups. First group : extubation is realised with aspiration in tracheal tube during removal tube Second group : extubation is realised without aspiration but with APL valve set to 20cmH20 Third group : extubation is realised without aspiration but with ventilator parameters were set for PSV mode (inspiratory pressure of 10cmH2O and PEEP identical to that administered in the operating room

ELIGIBILITY:
Inclusion Criteria:

* Visceral or urological surgery
* Scheduled surgery
* Surgical or patient requirement: placement of an arterial catheter
* Supine position
* Post-surgical extubation scheduled in the operating room
* Minimum age of 18 years
* Informed and signed consent

Exclusion Criteria:

* Severe obesity (BMI over 35kg/m2)
* pregnant woman
* Acute or chronic preoperative respiratory pathology.
* Sleep apnea syndrome
* Inability to receive informed information (does not speak, read or understand French)
* Patient under guardianship or curatorship
* Lack of social security coverage
* History of intubation or criteria for difficult intubation or ventilation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2022-06-29 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
desaturations during extubation | 1 minute after extubation
  saturation <92%

SECONDARY OUTCOMES:
desaturation postoperatory | 5 and 30 minutes after extubation
  saturation<92%
hypoxemia post operatory | 1 and 30 minutes after extubation
  PaO2 <60mmHg
atelectasis | 30 minutes after extubation
  Lung ultrasound score (LUS); min = 0, max = 32, higher scores mean is worse outcome
awakening time | through extubation completion, an average 2 minutes
  time in seconds
use of oxygen | day 7
  days Numbers of oxygen therapy, kinesiotherapy, non invasive ventilation
post operative complications | day 7 and day 28
  Clavien Dindo Score; min = grade I, max = grade V; higher scores mean is worse outcome
feasibility and acceptance of both techniques pressure positive extubation | 15 minutes after extubation
  questionnaire, min = 4, max =20, higher scores mean is worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Cédric CIRENEI, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Claude Huriez Chu Lille, Lille, France